CLINICAL TRIAL: NCT00658372
Title: A Phase 3, Randomized, Double-Blind, Parallel Group, 10-Week Placebo Controlled Fixed Dose Study Of PD 0332334 And Paroxetine Evaluating The Efficacy And Safety Of PD 0332334 For The Treatment Of Generalized Anxiety Disorder
Brief Title: A 10-week Study Evaluating the Efficacy and Safety of PD 0332334 in Patients With Generalized Anxiety Disorder (2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5361018
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: PD 0332334 phase 3 pivotal trial
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PD 0332334 225 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- PD 0332334 300 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- Paroxetine 20 mg QD (Active Comparator)
  Interventions: Drug: Paroxetine
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD 0332334 — Capsules, oral, 225 mg BID, 8 weeks with 2 week taper
  Other Names: imagabalin
  Arms: PD 0332334 225 mg BID
Drug: PD 0332334 — Capsules, oral, 300 mg BID, 8 weeks with 2 week taper
  Arms: PD 0332334 300 mg BID
Drug: Paroxetine — Capsules, oral, Paroxetine, 20 mg QD, 8 weeks with 2 week taper
  Arms: Paroxetine 20 mg QD
Drug: Placebo — Capsules, oral, placebo, BID, 8 weeks with 2 week taper
  Arms: Placebo BID

SUMMARY:
This is a 10-week trial that evaluates the efficacy and safety of PD 0332334 in subjects, ages 18 to 65, with generalized anxiety disorder.

DETAILED DESCRIPTION:
On February 23rd 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GAD (Diagnostic and Statistical Manual IV [DSM IV], 300.02) as established by the clinician (psychiatrist or licensed clinical psychologist) who has interviewed the subject using all sources of data including the Mini International Neuropsychiatric Interview (MINI) for DSM IV Axis I disorders and other clinical information. Subjects with specific phobia(s) (as defined in DSM IV) or dysthymic disorder will be allowed in the study.
* Subjects must have a HAM A total score ≥20 at the screening (V1) and randomization (V2) visits. Subjects must also have a Covi Anxiety Scale score of ≥9 and a Raskin Depression Scale score ≤7 at the Screening (V1) visit to ensure predominance of anxiety symptoms over depression symptoms.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, neurologic, active infections, immunological, or allergic disease (including drug allergies).
* Any of the following current (within the past 6 months through the present) DSM-IV Axis I diagnosis: Major Depressive Disorder, Obsessive Compulsive Disorder, Panic Disorder, Agoraphobia, Posttraumatic Stress Disorder, Anorexia, Bulimia, Caffeine induced anxiety disorder, Alcohol or substance abuse or dependence unless in full remission for at least 6 months, Social anxiety disorder.
* Any of the following past or current DSM-IV Axis I diagnoses: Schizophrenia, Psychotic disorder, Delirium, dementia, amnestic, and other clinically significant cognitive disorders, Bipolar or schizoaffective disorder, Cyclothymic disorder, Dissociative disorders.
* Antisocial or borderline personality disorder.
* Serious suicidal risk per the clinical investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The efficacy of PD 0332334 in the treatment of GAD will be measured by the change in the Hamilton Anxiety Rating Scale (HAM-A) total scores from baseline observed following 8 weeks of double-blind treatment. | 8 weeks
The safety and tolerability of PD 0332334 in subjects with GAD will be monitored in this study | 8 weeks

SECONDARY OUTCOMES:
Average (across the week 1, 2, 4, 6 and 8 visits) HAM-A change from baseline score | 8 weeks
Change from baseline in the HAM-A total score at weeks 1, 2, 4, and 6 | 6 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study Sleep Scale subscales | 8 weeks
Response rate on the patient-rated PGI-C at week 8 | 8 weeks
The "Week 1 Sustained Responder" rate based on the HAM A (where "Week 1 Sustained Responders" are defined as subjects with a 50% or greater improvement from baseline on the HAM A total score at Week 1 that is sustained until the Week 8 visit) | 1 week
Change from Baseline to Days 2- 8 and Weeks 2, 4, 6, 8 on the DAS A (total score) | 8 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study Sleep Scale (MOS SS) Sleep Disturbance Score | 8 weeks
Response rate on the HAM-A at week 1 and week 8 | 8 weeks
Change from Baseline to Week 1 on the Medical Outcomes Study Sleep Scale (MOS SS) Sleep Disturbance Score | 1 week
Change from baseline in the 17-item HAM-D total score at weeks 1, 2, 4, and 8 | 8 weeks
Change from Baseline in the psychic subscale score of the HAM A (Items 1- 6 and 14) at Week 8 | 8 weeks
Change from baseline in the somatic subscale score of the HAM-A (items 7 - 13) | 8 weeks
Change from baseline to week 8 in the QLesQ General Activity Score | 8 weeks
Worsening and improvement from baseline to week 8 on the changes in the Sexual Functioning Questionnaire (CSFQ) | 8 weeks
Remission rate based on the HAM A at Week 8 | 8 weeks
Response rate on the clinician-rated CGI-I ate week 1 and week 8 | 8 weeks
Change from baseline in CGI-S at week 8 | 8 weeks
Change from baseline to Days 2-8 and weeks 2, 4, 6 and 8 on the GA-VAS (diary) | 8 weeks
Change from baseline to week 8 on the Sheehan Disability Scale (SDS) total score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (28):
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Haverhill, Massachusetts
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
- Pfizer Investigational Site, Budapest, Hungary
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Tainan, Taiwan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361018&StudyName=A%2010-week%20study%20evaluating%20the%20efficacy%20and%20safety%20of%20PD%200332334%20in%20patients%20with%20generalized%20anxiety%20disorder%20%282%29